CLINICAL TRIAL: NCT07099937
Title: Metabolic Syndrome and Thyroid Dysfunction in Type 2 Diabetes In Upper Egypt
Brief Title: Relationship Between Thyroid Dysfunction and Diabetes
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ghada Ragab Hamed Abdelnasser, doctor, Assiut University
Other Study IDs: thyroid and diabetes mellitus
Record Dates: First submitted 2025-07-18; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Type 2 Diabetes Mellitus (T2DM); Thyroid Dysfunction; Metabolic Syndrome; Upper Egypt Patients
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational cross-sectional study with no intervention. — This study does not involve any intervention. It is a cross-sectional observational study. The term "intervention" here refers to laboratory investigations and clinical assessments conducted as part of data collection only.

SUMMARY:
Evaluate the expression of glycemic parameters, lipid profile, and thyroid hormones in patients with type 2 diabetes mellitus in upper egypt.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (T2DM) is a chronic metabolic disorder characterized by insulin resistance and impaired insulin secretion, resulting in persistent hyperglycemia. ( )..In T2DM, the response to insulin is diminished, and this is defined as insulin resistance. During this state, insulin is ineffective and is initially countered by an increase in insulin production to maintain glucose homeostasis, but over time, insulin production decreases, resulting in T2DM.( ).

Glycemic parameters are critical indicators for diagnosing and monitoring diabetes mellitus. The most commonly used measures include fasting blood glucose (FBG), postprandial blood glucose (PPBG), and glycated hemoglobin (HbA1c). Among them, HbA1c reflects the average blood glucose levels over the previous two to three months and is considered a reliable marker of chronic hyperglycemia.( ) Diabetic dyslipidemia constitutes a distinct cluster of plasma lipid and lipoprotein abnormalities that are metabolically interconnected in individuals with type 2 diabetes mellitus. This condition is predominantly characterized by elevated triglyceride (TG) concentrations, reduced levels of high-density lipoprotein cholesterol (HDL-C) ( ).

The underlying mechanism involves insulin resistance, which disrupts normal lipid metabolism by enhancing hepatic very low-density lipoprotein (VLDL) synthesis and impairing the clearance of triglyceride-rich lipoproteins. ( ) Prevalence of thyroid dysfunction is greater in diabetes patients compared to the general population.1-3 Prevalence of thyroid dysfunction in general population is around 6.6-13.4%, while in diabetes population around 10-24%.1 Studies found that subclinical hypothyroidism is the most common thyroid dysfunction in diabetic population ( ) Emerging evidence suggests a complex interplay between glycemic control, lipid metabolism, and thyroid function in patients with type 2 diabetes mellitus. Poor glycemic control has been associated with adverse lipid profiles and alterations in thyroid hormone levels, which may collectively contribute to the progression of diabetic complications. Thyroid hormones influence both glucose and lipid metabolism by regulating hepatic glucose production, lipolysis, and insulin sensitivity. ( ).

This study was conducted in Upper Egypt, a region characterized by distinct sociodemographic and health profiles compared to other parts of the country. Despite the growing burden of non-communicable diseases, including type 2 diabetes, there is a noticeable lack of regional epidemiological data addressing the coexistence of metabolic syndrome and thyroid dysfunction. Investigating this relationship in the Upper Egypt population may help fill existing knowledge gaps and support the development of more effective, geographically tailored healthcare strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with type 2 diabetes mellitus in upper egypt.
* Age above 18 years.
* Patients who gave informed consent to participate.

Exclusion Criteria:

* Patients with type 1 diabetes mellitus.
* Age below 18 years.
* Patients with known autoimmune thyroid diseases, pregnancy, or acute illness at the time of assessment.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 18 years and above diagnosed with type 2 diabetes mellitus attending the Diabetes and Endocrinology Outpatient Clinic at Assiut University Hospitals, Upper Egypt.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Prevalence of thyroid dysfunction among type 2 diabetic patients | Baseline
  The outcome will measure the proportion (%) of type 2 diabetic patients diagnosed with thyroid dysfunction. This includes classification into hypothyroidism, hyperthyroidism, subclinical hypothyroidism, and subclinical hyperthyroidism based on standard laboratory cutoffs of TSH, free T3, and free T4.
Association between thyroid dysfunction and metabolic syndrome in type 2 diabetic patients | Baseline
  The outcome will assess the statistical correlation (e.g., chi-square test or logistic regression) between the presence of thyroid dysfunction and the diagnosis of metabolic syndrome, according to IDF criteria. Results will be reported as odds ratios or p-values as appropriate.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sakamoto M. Type 2 Diabetes and Glycemic Variability: Various Parameters in Clinical Practice. J Clin Med Res. 2018 Oct;10(10):737-742. doi: 10.14740/jocmr3556w. Epub 2018 Sep 10. PMID 30214644
- [Background] Ford ES, Li C, Sattar N. Metabolic syndrome and incident diabetes: current state of the evidence. Diabetes Care. 2008 Sep;31(9):1898-904. doi: 10.2337/dc08-0423. Epub 2008 Jun 30. PMID 18591398
- [Background] Hadgu R, Worede A, Ambachew S. Prevalence of thyroid dysfunction and associated factors among adult type 2 diabetes mellitus patients, 2000-2022: a systematic review and meta-analysis. Syst Rev. 2024 Apr 30;13(1):119. doi: 10.1186/s13643-024-02527-y. PMID 38689302
- [Background] Chen H, Wu J, Lyu R. Expressions of glycemic parameters, lipid profile, and thyroid hormone in patients with type 2 diabetes mellitus and their correlation. Immun Inflamm Dis. 2024 Jul;12(7):e1282. doi: 10.1002/iid3.1282. PMID 38967365